CLINICAL TRIAL: NCT06328127
Title: Positive Psychology Intervention for Hematopoietic Stem Cell Transplantation Survivors
Acronym: PATH-4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Duke University (Other); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Principal Investigator, Hermioni L.Amonoo, MD, MPP, MPH, Director, Well-Being and Cancer Research Program, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-691
Record Dates: First submitted 2024-03-11; First posted 2024-03-25 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: stem cell transplant; positive psychology intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Affect in the Transplantation of Hematopoietic Stem Cells (PATH) (Experimental): Participants recruited from the Dana-Farber Cancer Institute, Duke Cancer Institute, and Moffitt Cancer Center who are randomized to the intervention/experimental arm will receive the PATH intervention, which is focused on gratitude, strengths, and meaning, as well as focused exercises on goal-setting and tracking daily physical activity.
  Participants will complete questionnaires (in person, over the computer or telephone, or by mail) at predetermined days per protocol.
  Interventions: Behavioral: PATH
- Usual Care (No Intervention): Participants recruited from the Dana-Farber Cancer Institute, Duke Cancer Institute, and Moffitt Cancer Center who are randomized to the usual care arm will receive their usual support from the HSCT team, including all routine supportive care resources (e.g., support from social work) offered by the HSCT team.
  Participants will complete questionnaires (in person, over the computer or telephone, or by mail) at predetermined days per protocol.

INTERVENTIONS:
Behavioral: PATH — PATH, a phone-delivered positive psychology intervention for patients who have undergone HSCT, consists of three 3-week modules. The first module focuses on gratitude and physical activity goal setting. The second module focuses on personal strengths and resources to enhance daily physical activity. The third module focuses on meaning and assessing barriers to physical activity. The third week of each module is an integration exercise dedicated to help participants explore practical ways of incorporating the themes for the given module into daily life. A trained interventionist will guide participants to complete each 30-minute weekly session.
  Arms: Positive Affect in the Transplantation of Hematopoietic Stem Cells (PATH)

SUMMARY:
This randomized clinical trial is evaluating the impact of a positive psychology intervention (PATH) on anxiety symptoms, depression symptoms, and quality of life in survivors of hematopoietic stem cell transplant (HSCT) compared to usual care.

DETAILED DESCRIPTION:
Patients undergoing hematopoietic stem cell transplantation (HSCT) deal with numerous physical and psychological symptoms during acute hospitalization and recovery. Of the few psychosocial interventions tailored to the needs of the HSCT population, most focus on the needs of patients in the pre-transplant phase or during the HSCT hospitalization, but not during the acute recovery period starting at 100-days post-HSCT. Hence, the investigators developed a remotely-delivered positive psychology intervention, Positive Affect in the Transplantation of Hematopoietic Stem Cells (PATH). This intervention encourages patients to perform simple and enjoyable structured activities that increase the intensity of positive thoughts and emotions. With this multi-site randomized clinical trial, the investigators aim to find out whether PATH can improve psychological distress and quality of life in HSCT survivors, compared to usual care, using validated assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years and older) undergoing allogeneic HSCT and are approaching 100-days post-HSCT
* Ability to speak, read, and respond to questions in English or Spanish to complete study procedures
* Access to a basic telephone

Exclusion Criteria:

* Patients who underwent allogeneic HSCT for benign hematologic conditions
* Patients with severe psychiatric or cognitive conditions, such as dementia, determined by their transplant oncologist to make them unable to provide informed consent or comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety Symptoms based on the Hospital Anxiety and Depression Scale-Anxiety Subscale | 10 weeks
  Compare anxiety symptoms between the two groups at 10 weeks using the 7-item Hospital Anxiety and Depression Scale-Anxiety subscale (HADS-A).
  The HADS-A subscale ranges from 0-21, with higher scores indicating worse anxiety symptoms.

SECONDARY OUTCOMES:
Anxiety Symptoms based on the Hospital Anxiety and Depression Scale-Anxiety Subscale | Up to 40 weeks
  Compare anxiety symptoms longitudinally between the two groups using the 7-item Hospital Anxiety and Depression Scale-Anxiety (HADS-A) subscale.
  The HADS-A subscale ranges from 0-21, with higher scores indicating worse anxiety symptoms.
Depression Symptoms based on the Hospital Anxiety and Depression Scale-Depression Subscale | Up to 40 weeks
  Compare depression symptoms longitudinally between the two groups using the 7-item Hospital Anxiety and Depression Scale-Depression (HADS-D) subscale.
  The HADS-D subscale ranges from 0-21, with higher scores indicating worse depression symptoms.
Gratitude based on the Gratitude Questionnaire | Up to 40 weeks
  Compare gratitude longitudinally between the two groups using the 6-item Gratitude Questionnaire.
  The Gratitude Questionnaire ranges from 6-42, with higher scores indicating a stronger propensity for experiencing gratitude in daily life.
Positive Affect based on the Positive and Negative Affect Schedule Positive Affect Subscale | Up to 40 weeks
  Compare positive affect longitudinally between the two groups using the 10-item Positive and Negative Affect Schedule (PANAS) Positive Affect Subscale.
  The PANAS Positive Affect Subscale ranges from 10-50, with higher scores indicating higher levels of positive affect.
Physical function based on the Patient-Reported Outcomes Measurement Information System-Physical Function-20 | Up to 40 weeks
  Compare physical function longitudinally between the two groups using the 20-item Patient-Reported Outcomes Measurement Information System-Physical Function-20 (PROMIS-PF-20).
  The PROMIS-PF-20 ranges from 20 to 100, with higher scores indicating better physical functioning.
Patient-Reported Quality of Life based on the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) | Up to 40 weeks
  Compare quality of life longitudinally between the two groups using the 47-item Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT).
  The FACT-BMT consists of 5 subscales assessing well-being across the following domains: physical, functional, emotional, social, and bone marrow transplant symptoms. The FACT-BMT ranges from 0-148, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hermioni Amonoo, MD, MPP, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Cancer Institute, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber/Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor, Investigator, or designee. The protocol and statistical analysis plan will be made available on ClinicalTrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the study investigator at hermioni_amonoo@dfci.harvard.edu